CLINICAL TRIAL: NCT05958459
Title: The Effect of Eye Exercises for the Stimulation of Neuroadaptation After Multifocal Intraocular Lens Implantation on Visual Function and Quality of Life
Brief Title: The Effect of Eye Exercises on Visual Function and Quality of Life After Multifocal Intraocular Lens Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Idrıs Dogan (Other)
Responsible Party: Sponsor-Investigator, Idrıs Dogan, lecturer, Batman University
Organization: Batman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-DOGAN-001
Record Dates: First submitted 2023-07-05; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Cataract; Intraocular Lenses
Keywords: Cataract; Eye Exercises; Neuroadaptation; Intraocular Lens; Life quality; visual function
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): The individuals in the study group will perform home-based eye exercises for at least 1 session (~30 min.) every day for a total of 12 weeks, after the patient's condition is stable, starting from the 7th day after the surgery. After the initial assessment, participants will be given illustrated brochures describing the exercises and will be taught how to perform the exercises. Whether individuals comply with the exercise program will be closely monitored (by keeping a diary, online meetings and periodically calling individuals). Eye exercises include eight steps. These; Covering the eyes with the palm of the hand, blinking, lateral gaze, anterior and lateral gaze, rotational gaze, up-down gaze, nasal tip gaze, and near and far gaze.
  Interventions: Other: Eye Exercise
- control group (Experimental): The control group, on the other hand, will not perform any exercise, but will only be evaluated.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: Eye Exercise — The individuals in the study group will perform home-based eye exercises for at least 1 session (~30 min.) every day for a total of 12 weeks, after the patient's condition is stable, starting from the 7th day after the surgery. After the initial assessment, participants will be given illustrated brochures describing the exercises and will be taught how to perform the exercises. Whether individuals comply with the exercise program will be closely monitored (by keeping a diary, online meetings and periodically calling individuals). The control group, on the other hand, will not perform any exercise, but will only be evaluated. Eye exercises include eight steps. These; Covering the eyes with the palm of the hand, blinking, lateral gaze, anterior and lateral gaze, rotational gaze, up-down gaze, nasal tip gaze, and near and far gaze.
  Arms: study group
Other: no intervention — no intervention
  Arms: control group

SUMMARY:
The goal of this clinical trial is to examine the effects of eye exercises on visual function and quality of life in cataract patients undergoing multifocal intraocular lens implantation. The main questions it aims to answer are:

* Does it improve visual functions?
* Does it improve vision-related quality of life?

Participants in the intervention group will perform 8-step eye exercises at least once a day for 12 weeks. The control group will not practice, they will only be evaluated.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial to be performed on individuals implanted with multifocal intraocular lenses. Necessary permissions were obtained from Hasan Kalyoncu University Non-Interventional Research Ethics Committee, Private Batman Dunya and Private Batman MedicalPoint Hospitals for the study. Participants will be selected from patients who are scheduled for multifocal intraocular lens implantation in the ophthalmology units of the relevant hospitals, who agree to volunteer and sign an informed consent form.

The individuals participating in the study will be randomly divided into two groups as the study group and the control group. Participants will be evaluated for a total of 3 times: before the surgery, at the 1st and 3rd months after the surgery. The number of group participants will be determined according to the power analysis of the data obtained in the first evaluation and considering data loss.

DATA TO BE COLLECTED:

* Demographic information (name, surname, contact information, age, weight, height, occupation, education level, CV, family history, medication, etc.),
* Refractive errors (Astigmatism, myopia, etc.),
* Near, medium, far visual acuity (Snellen Chart),
* Contrast sensitivity (Pelli-Robson contrast sensitivity chart),
* Pupillary Diameter,
* Intraocular pressure,
* Reading speed,
* Vision-related quality of life (National Institute of Eye Health Visual Function Scale (NEI-VFQ-25),
* Anxiety level (State and Trait Anxiety Scale),
* Cognitive performance (Standardized Mini Mental Test).

Refraction errors, visual acuity (near, intermediate and far), contrast sensitivity, intraocular pressure and pupil diameter will be evaluated by the ophthalmologist.

The individuals in the study group will perform home-based eye exercises for at least 1 session (~30 min.) every day for a total of 12 weeks, after the patient's condition is stable, starting from the 7th day after the surgery. After the initial assessment, participants will be given illustrated brochures describing the exercises and will be taught how to perform the exercises. Whether individuals comply with the exercise program will be closely monitored (by keeping a diary, online meetings and periodically calling individuals). The control group, on the other hand, will not perform any exercise, but will only be evaluated. Eye exercises include eight steps. These; Covering the eyes with the palm of the hand, blinking, lateral gaze, anterior and lateral gaze, rotational gaze, up-down gaze, nasal tip gaze, and near and far gaze.

* Closing the eyes with the palms; It helps to correct visual defects by stimulating eye muscles and stimulating aqueous humor circulation.
* Blinking; It supports the spontaneous realization of eye reflexes and helps to relax the eye muscles.
* sideways view; It relieves the tension of the eye muscles caused by close work and continuous reading and helps to correct strabismus.
* Front and side view; It regulates the coordination of the medial and lateral eye muscles.
* rotational view; regulates the balance of coordinated and peripheral movements of each eyeball.
* Up and down view; Balances the upper and lower eye muscles.
* Looking at the tip of the nose; It helps to focus the eye muscles and provide accommodation.
* Finally, the near and far gaze is similar to the nose tip, but the range of motion is wider.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who can read,
* To adapt to the training program,
* To be involved in working voluntarily,

Exclusion Criteria:

* Individuals with a history of eye surgery,
* Being diagnosed with strabismus,
* Being diagnosed with glaucoma,
* Having a history of neurological disease that will affect vision and eye muscles,
* Having retinal and visual pathway damage,
* Having functional damage that will prevent the practice of exercises.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-04 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Contrast Sensitivity | 12 Week (3 times in total, before the operation, at the 1st and 3rd months after the operation.)
  The Pelli-Robson contrast sensitivity test is a wall chart measuring 90 X 60 cm. The chart comprises 8 lines of letters with different contrasts. Each line has 6 letters; the first 3 letters (a triplet) on the left have more contrast than the 3 letters on the right. The contrast also decreases downward from line to line. The size of the letters is 4.9 X 4.9 cm. There are different sets of letters on each side of the chart. It recommends a test distance of 1 m. The logarithmic contrast sensitivity value of the last triplet of which at least 2 letters are correctly seen is marked as the result. The luminance of the test should be 85 candelas/m2 (cd/m2 ); the accepted range is 60 to 120 cd/m2.
Visual acuity | 12 Week (3 times in total, before the operation, at the 1st and 3rd months after the operation.)
  Snellen chart will be used for visual acuity measurement.
Vision-related quality of life | 12 Week (3 times in total, before the operation, at the 1st and 3rd months after the operation.)
  The National Institute of Eye Health Visual Function Scale (NEI-VFQ-25) will be used. This scale is used to evaluate visual function loss due to eye diseases and was developed by Mangione et al. in 1988. In order to make this scale, whose original form consists of 51 questions, more useful, a 25-question form was developed. The short form of 25 questions consists of 3 parts. These sections are respectively; general health and vision, difficulties with activities, and the consequences of vision problems.

SECONDARY OUTCOMES:
Refraction errors | 12 Week (3 times in total, before the operation, at the 1st and 3rd months after the operation.)
  The refraction defects were measured by autorefractometry, which is frequently used because it provides fast and reliable results in clinic. In the autorefractometry method, the infrared rays sent to the patient's eye are reflected from the retina back to the device and evaluate the refraction defect of the patient
İntraocular Pressure | 12 Week (3 times in total, before the operation, at the 1st and 3rd months after the operation.)
  It will be measured with the Reichert 7CR Automatic Non Contact Tonometer device.
Pupillary diameter | 12 Week (3 times in total, before the operation, at the 1st and 3rd months after the operation.)
  will be evaluated using optical biometry.
Reading speed | 12 Week (3 times in total, before the operation, at the 1st and 3rd months after the operation.)
  Written material prepared in Times New Roman font and 12 point size will be read to the participant for one minute under appropriate lighting. At the end of the one-minute reading period, correctly read and incorrectly read words will be counted. The numerical value obtained by subtracting the number of words read incorrectly from the number of words read correctly will be used as a measure of the participant's reading speed.

OTHER OUTCOMES:
Demographic information | Only on the first assessment (through study completion, an average of 12 week)
  name, surname, contact information, age, weight, height, occupation, education level, CV, family history, medication, etc.
anxiety level (State Trait Anxiety Inventory I-II) | 12 Week (3 times in total, before the operation, at the 1st and 3rd months after the operation.)
  The response options collected in four classes in the state anxiety scale are (1) Not at all, (2) A little, (3) A lot, and (4) Completely; The options in the Trait Anxiety Scale are (1) Almost never, (2) Sometimes, (3) Often, and (4) Almost always. There are two kinds of expressions in the scales. We can call these (1) direct or straight statements and (2) inverted statements. Direct expressions, negative emotions; reversed expressions express positive emotions. When scoring this second type of statements, those with a weight of 1 turn into 4, and those with a weight of 4 turn into 1. In direct statements, answers with a value of 4 indicate high anxiety. In reversed statements, answers with a value of 1 indicate high anxiety, and those with a value of 4 indicate low anxiety. The scores obtained from both scales theoretically vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
cognitive performance | Only on the first assessment (through study completion, an average of 12 week)
  Standardized Mini Mental Test will be used.